CLINICAL TRIAL: NCT00000644
Title: A Phase II Safety and Efficacy Study of Clarithromycin in the Treatment of Disseminated M. Avium Complex (MAC) Infections in Patients With AIDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Abbott (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 157
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Mycobacterium Avium-intracellulare Infection; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Mycobacterium avium-intracellulare Infection; Acquired Immunodeficiency Syndrome; Clarithromycin
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Clarithromycin

INTERVENTIONS:
Drug: Clarithromycin

SUMMARY:
This study is designed to evaluate the efficacy and safety of clarithromycin given orally at 1 of 3 doses to treat disseminated Mycobacterium avium complex infections (MAC) in patients with AIDS.

Mycobacterium avium complex (MAC) is thought to be the most common disseminated bacterial opportunistic infection in AIDS, with clinical prevalence estimates ranging from 15 to 50 percent of all AIDS patients. Clarithromycin, a new macrolide antimicrobial agent, has demonstrated activity against MAC both in the laboratory and in animals. Clinical experience treating AIDS patients with clarithromycin for disseminated MAC is limited. However, early studies have indicated few adverse effects and some improvement in clinical symptoms scores and Karnofsky performance scores over placebo treated patients.

DETAILED DESCRIPTION:
Mycobacterium avium complex (MAC) is thought to be the most common disseminated bacterial opportunistic infection in AIDS, with clinical prevalence estimates ranging from 15 to 50 percent of all AIDS patients. Clarithromycin, a new macrolide antimicrobial agent, has demonstrated activity against MAC both in the laboratory and in animals. Clinical experience treating AIDS patients with clarithromycin for disseminated MAC is limited. However, early studies have indicated few adverse effects and some improvement in clinical symptoms scores and Karnofsky performance scores over placebo treated patients.

Treatment is randomly assigned so that twice as many patients receive clarithromycin at the lower dose as at an intermediate dose for 12 weeks. Once data becomes available to support dosing patients with clarithromycin at the highest dose, then treatment will be randomly assigned so that twice as many patients receive clarithromycin at the highest dose as at the intermediate dose. Sixteen patients per group (48 patients in all) will be enrolled. Patients exhibiting clinical improvement or clinical cure while on this trial will be allowed to continue on therapy for an additional 6 months. Patients will have clinical evaluations (including the Karnofsky Performance Scale), laboratory evaluations (hematology and chemistry), and blood cultures for MAC performed monthly.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Didanosine (ddI).
* Dideoxycytidine (ddC).
* Zidovudine (AZT).
* Acetaminophen.
* Acyclovir.
* Fluconazole.
* Erythropoietin (EPO).
* Systemic Pneumocystis carinii pneumonia (PCP) prophylaxis (aerosolized or oral pentamidine, trimethoprim / sulfamethoxazole, or dapsone).
* Maintenance ganciclovir therapy (permitted only if dose and clinical and laboratory parameters have been stable for at least 4 weeks prior to study entry).
* Maintenance treatment for other opportunistic infections if the dose and clinical and laboratory parameters have been stable for 4 weeks prior to study entry.

Patients must have:

* Positive results for HIV by ELISA confirmed by another method.
* Positive blood culture for Mycobacterium avium complex within 2 months of study entry and clinical symptoms of MAC infection.
* Discontinued all mycobacterial drugs (approved and investigational) for at least 4 weeks prior to the start of drug therapy (with the exception of isoniazid prophylaxis which should be discontinued at Study Day minus 14 to Study Day minus 7
* Given written informed consent to participate in the trial.
* Met the listed laboratory parameters in the pre-treatment visit.

Prior Medication:

Allowed:

* Didanosine (ddI).
* Deoxycytidine (ddC).
* Zidovudine (AZT).
* Acetaminophen.
* Acyclovir.
* Fluconazole.
* Erythropoietin (EPO).
* Systemic Pneumocystis carinii pneumonia (PCP) prophylaxis (aerosolized or oral pentamidine, dapsone, trimethoprim / sulfamethoxazole).
* Maintenance ganciclovir therapy (permitted only if dose and clinical and laboratory parameters have been stable for at least 4 weeks prior to study entry).

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Active opportunistic infections. Maintenance treatment for other opportunistic infections will be permitted if the dose and clinical and laboratory parameters have been stable for 4 weeks prior to study entry.

Concurrent Medication:

Excluded:

* Aminoglycosides.
* Ansamycin (rifabutin).
* Quinolones.
* Other macrolides.
* Clofazimine.
* Cytotoxic chemotherapy.
* Rifampin.
* Ethambutol.
* Immunomodulators (except alpha interferon).
* Investigational drugs (except ddI, ddC, and erythropoietin).

Patients with the following are excluded:

* History of allergy to macrolide antimicrobials.
* Currently on active therapy with any anti-mycobacterial drugs listed in Exclusion Prior Medications.
* Currently on active therapy with carbamazepine or theophylline, unless the investigator agrees to carefully monitor blood levels.
* Inability to comply with the protocol or judged to be near imminent death by the investigator.
* Active opportunistic infections.
* Requiring any of the excluded concomitant medications.

Prior Medication:

Excluded for at least 4 weeks prior to study entry:

* All anti-mycobacterial drugs (approved and investigational) with the exception of isoniazid prophylaxis, which should be discontinued at Study Day minus 14 to minus 7.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Primary Completion 1997-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chaisson R, Study Chair
Locations (3):
- United States (3):
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Johns Hopkins Hosp, Baltimore, Maryland

REFERENCES:
- [Background] Chaisson RE, Benson CA, Dube MP, Heifets LB, Korvick JA, Elkin S, Smith T, Craft JC, Sattler FR. Clarithromycin therapy for bacteremic Mycobacterium avium complex disease. A randomized, double-blind, dose-ranging study in patients with AIDS. AIDS Clinical Trials Group Protocol 157 Study Team. Ann Intern Med. 1994 Dec 15;121(12):905-11. doi: 10.7326/0003-4819-121-12-199412150-00001. PMID 7978715
- [Background] Wu AW, Lichter SL, Richardson W, Urbanski PA, Benson C, Sattler FR, Chaisson R. Quality of life in patients receiving clarithromycin for Mycobacterium avium complex infection and AIDS. Int Conf AIDS. 1992 Jul 19-24;8(2):B178 (abstract no PoB 3550)
- [Background] Chaisson RE, Benson CA, Dube M, Hafner R, Dellerson M, Lichter S, Smith T, Sattler FR. Clarithromycin for disseminated Mycobacterium avium-complex in AIDS patients. Int Conf AIDS. 1992 Jul 19-24;8(1):We54 (abstract no WeB 1052)